CLINICAL TRIAL: NCT05388513
Title: Evaluating Factors Affecting Survival in Colon and Rectum Cancer: A Prospective Cohort Study With 161 Patients
Brief Title: Evaluating Factors Affecting Survival in Colon and Rectum Cancer
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Fatih Basak, Clinical Associate Professor, Umraniye Education and Research Hospital
Other Study IDs: ColoRectalCancers
Record Dates: First submitted 2016-09-07; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Colon Cancer; Rectum Cancer
Keywords: Survival; Prognostic factors
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colon: The patients who are operated with colon cancer
  Interventions: Procedure: Surgical Resection
- Rectum: The patients who are operated with rectum cancer
  Interventions: Procedure: Surgical Resection

INTERVENTIONS:
Procedure: Surgical Resection — Surgically treated patients included

SUMMARY:
Colorectal cancers are frequent among cancers of the gastrointestinal system. Whether there are any differences between survival in rectum and colon cancer patients is controversial. This study aimed to compare survival in the surgically treated rectum and colon cancers and determine the factors affecting survival.

DETAILED DESCRIPTION:
Colorectal cancers are frequent in the gastrointestinal system. It is the 4th most common cancer after lung, prostate, and bladder in the male population and it is the 3rd after breast and thyroid cancers in the female population according to World Health Organization. It is considered significant morbidity and mortality cause and is estimated to develop in more than 1.000.000 individuals annually worldwide. Colorectal cancers form 10% of all cancers in the female and male populations. It is the 2nd most common cause of death among cancers in the United States of America.

In studies, it is stated that the risk of developing colorectal cancer in an individual is 5-6%. Also, the risk of death of an individual due to colorectal cancer was determined as 3%. In the last 50 years, the rate of colorectal cancer mortality decreased in the female population while it did not change in the male population. Whether there is a difference in survival time between rectum and colon cancers is controversial.

With the development in neoadjuvant treatment approaches, poor prognosis in past years got better. Recent studies show that the prognosis in rectum cancers is better than in colon. Nevertheless, factors affecting prognosis other than treatment for both colon and rectum cancers are not clarified.

In this study, the investigators aimed to evaluate the surgically treated rectum and colon cancer patients' survival and factors affecting survival time.

ELIGIBILITY:
Inclusion Criteria:

Patients who were operated and diagnosed histopathologically as adenocarcinoma were included.

Exclusion Criteria:

Inoperable and recurrent colorectal cancer patients and patients that were diagnosed with other than adenocarcinoma were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients with colon and rectum cancer operated were examined
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Survival | 5 year
  5 year survival data is used.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Başak, Principal Investigator — Umraniye Education and Research Hospital

IPD SHARING:
Plan to Share IPD: No